CLINICAL TRIAL: NCT05594147
Title: COVID-19 Related Outcomes Among Cancer Patients Treated With TKIs, Including RegorafeNib or SorAfenib
Brief Title: An Observational Study, Called ROCURS, to Learn About COVID-19 Related Outcomes in People With Cancer Who Are Treated With Tyrosine Kinase Inhibitors (TKIs) Including Regorafenib or Sorafenib
Acronym: ROCURS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22294
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Malignant Solid Tumors; Coronavirus Disease 2019 (COVID-19); SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — regorafenib; Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TKIs treated group: Adult cancer patients with newly diagnosed COVID-19 who used Tyrosine kinase inhibitors (TKIs) within 30 days before COVID-19 diagnosis.
  Interventions: Drug: Other TKIs; Drug: Regorafenib (Stivarga, BAY73- 4506); Drug: Sorafenib (Nexavar, BAY43-9006)
- Non-TKIs treated group: Adult cancer patients with newly diagnosed COVID-19 who used other anti-cancer therapies 30 days before COVID-19 diagnosis
  Interventions: Drug: Non-TKIs

INTERVENTIONS:
Drug: Non-TKIs — Retrospective cohort analysis, using IBM MarketScan and Optum Clinformatics database in the US.
  Groups: Non-TKIs treated group
Drug: Other TKIs — Retrospective cohort analysis, using IBM MarketScan and Optum Clinformatics database in the US.
  Groups: TKIs treated group
Drug: Regorafenib (Stivarga, BAY73- 4506) — Retrospective cohort analysis, using IBM MarketScan and Optum Clinformatics database in the US.
  Groups: TKIs treated group
Drug: Sorafenib (Nexavar, BAY43-9006) — Retrospective cohort analysis, using IBM MarketScan and Optum Clinformatics database in the US.
  Groups: TKIs treated group

SUMMARY:
This is an observational study in which data from people with cancer who had the Coronavirus disease 2019 (COVID-19) are collected and studied. In observational studies, only observations are made without specified advice or interventions.

The most recently discovered coronavirus (SARS-CoV-2) may cause illness in humans ranging from the common cold to serious illness, also known as COVID-19.

People with cancer are particularly at risk of becoming very sick with COVID-19, especially during or shortly after a cancer treatment. Several treatments for COVID-19 have been tested in clinical studies. However, people with cancer or with recent cancer treatments were usually excluded.

Tyrosine kinase inhibitors (TKIs) are used to treat several cancer types. TKIs including regorafenib and sorafenib block certain proteins, which are involved in the growth of cancer. They also have an anti-inflammatory effect and may be able to block the entry of the coronavirus into the cell. This could possibly prevent infection. However, data on COVID-19 from people with cancer receiving TKIs are missing.

The main purpose of this study is to find out whether COVID-19 outcomes were different in people with cancer receiving TKIs compared to those receiving other anti-cancer drugs. To do this, researchers will compare COVID-19 outcomes within 30 days of COVID-19 diagnosis between both groups.

The data for the comparison will come from databases called Optum and MarketScan.

Besides this data collection, no further tests or examinations are planned in this study.

There are no required visits or tests in this study. Data will be from October 2019 to June 2021 or the latest available data.

ELIGIBILITY:
Inclusion Criteria:

TKIs Treated Group

* Patients ≥18 years old at index date
* Patients who had any healthcare encounter with a primary or secondary diagnosis of Coronavirus disease 2019 (COVID-19) or positive results from Polymerase Chain Reaction (PCR) lab test for Severe acute respiratory syndrome coronavirus 2 (SARs-CoV-2) during the patient identification period (January 1, 2020 to May 31, 2021 or one month before the latest data cut)
* Patient who was under TKIs on index date or the last episode of TKIs treatment ended within 30 days before index date
* Patient who had any diagnosis of solid tumors at any time before index date (identified using ICD-9 or ICD-10 diagnosis codes, Supplementary Table 5)
* Continuous insurance enrollment for at least 90 days before index date

Non-TKIs Treated Group

* Patients ≥18 years old at index date
* Patients who had any healthcare encounter with a primary or secondary diagnosis of COVID-19 or positive results from PCR lab test for SARs-CoV-2 during the patient identification period
* Patient who had any diagnosis of solid tumors any time before the index
* Patient who was under anti-neoplastic medications on index date or the last episode of the anti-neoplastic treatment ended within 30 days before index date
* Continuous insurance enrollment for at least 90 days before index date

Exclusion Criteria:

TKIs treated Group

- Patients who had secondary cancer without site specification (only had ICD-10 codes C79.9 or C80 for metastasis) from 90 days before index

Non-TKIs Treated Group

* Patients who had any claims of TKIs treatment during the study period
* Patients who had secondary cancer without site specification (only had ICD-10 codes C79.9 or C80 for metastasis) from 90 days before index

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients with newly diagnosed COVID-19 (the first incidence of COVID-19) who were under TKIs therapy or within 30 days after the last TKIs therapy at the first incidence of COVID-19 from October 1, 2019 to June 30, 2021 or the latest data cut in the databases, will be included in the TKIs treated group. Similarly, newly diagnosed COVID-19 patients who did not receive any TKIs during the same study period will be selected in the non-TKIs treated group.
Sampling Method: Non-Probability Sample
Enrollment: 4103 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
All-cause mortality for TKI-treated group and non-TKI-treated group | Retrospective data analysis from October 2019 to June 2021
  This analysis will use subjects from Optum only.
COVID-19 related hospitalizations for TKI-treated group and non-TKI-treated group | Retrospective data analysis from October 2019 to June 2021
  Any inpatient visit with a diagnosis of COVID-19
Intensive Care Unit (ICU) admission during COVID-19 related hospitalization for TKI-treated group and non-TKI-treated group | Retrospective data analysis from October 2019 to June 2021
Use of mechanical ventilator during COVID-19 related hospitalization for TKI-treated group and non-TKI-treated group | Retrospective data analysis from October 2019 to June 2021
Emergency room visit with a diagnosis of COVID-19 for TKI-treated group and non-TKI-treated group | Retrospective data analysis from October 2019 to June 2021
Newly diagnosed COVID-19 related complications (not present at baseline) for TKI-treated group and non-TKI-treated group | Retrospective data analysis from October 2019 to June 2021
  Complications Including:
  1. Pneumonia
  2. Multisystem inflammatory syndrome
  3. Acute hepatic failure
  4. Acute kidney failure
  5. Acute myocarditis
  6. Acute respiratory distress syndrome
  7. Cardia arrhythmia
  8. Sepsis
  9. Viral cardiomyopathy
  10. Viral pericarditis

SECONDARY OUTCOMES:
All-cause mortality for Regorafenib or Sorafenib treated group and non-TKI-treated group | Retrospective data analysis from October 2019 to June 2021
COVID-19 related hospitalizations for Regorafenib or Sorafenib treated group and non-TKI-treated group | Retrospective data analysis from October 2019 to June 2021
Intensive Care Unit (ICU) admission during COVID-19 related hospitalization Regorafenib or Sorafenib treated group and non-TKI-treated group | Retrospective data analysis from October 2019 to June 2021
Use of mechanical ventilator during COVID-19 related hospitalization Regorafenib or Sorafenib treated group and non-TKI-treated group | Retrospective data analysis from October 2019 to June 2021
Emergency room visit with a diagnosis of COVID-19 Regorafenib or Sorafenib treated group and non-TKI-treated group | Retrospective data analysis from October 2019 to June 2021
Newly diagnosed COVID-19 related complications (not present at baseline) Regorafenib or Sorafenib treated group and non-TKI-treated group | Retrospective data analysis from October 2019 to June 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.